CLINICAL TRIAL: NCT05511662
Title: Influence of Patient-reported Outcome Follow-up Based on the Northern Shanghai Community Chronic Disease Management System on the Follow-up Compliance and Satisfaction of Patients With Atrial Fibrillation After Cryoablation.
Brief Title: Patient-reported Outcome Follow-up Based on the Northern Shanghai Community Chronic Disease Management System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director of Cardiology, Shanghai 10th People's Hospital
Other Study IDs: NSH-PRO
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; follow up；patient-reported outcomes；
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- routine follow-up: The patients were instructed to come to the hospital for routine follow-up at 1, 3, 6, and 12 months after the operation. If necessary, the investigators contacted the patients by phone for symptom follow-up and instructed them to come to the hospital for relevant examinations (eg: EKG, Holter, echocardiography, etc.)
- PRO follow-up: On the basis of the routine follow-up group, interactive follow-up was conducted through the chronic disease follow-up system, including the APP for regular follow-up (bound to sign the informed consent form, and the account of the patient and his immediate family who can be familiar with the WeChat applet), SMS reminders, and doctors when necessary. Wechat/platform communication and exchange, inappropriate ECG data upload and other multi-dimensional follow-up, at the same time assisting the ECG integrated follow-up platform for ECG data management and medication guidance.
  Interventions: Other: PRO follow up

INTERVENTIONS:
Other: PRO follow up — On the basis of the routine follow-up group, interactive follow-up was conducted through the chronic disease follow-up system, including the APP for regular follow-up (bound to sign the informed consent form, and the account of the patient and his immediate family who can be familiar with the WeChat applet), SMS reminders, and doctors when necessary. Wechat/platform communication and exchange, inappropriate ECG data upload and other multi-dimensional follow-up, at the same time assisting the ECG integrated follow-up platform for ECG data management and medication guidance
  Groups: PRO follow-up

SUMMARY:
Influence of patient-reported outcome follow-up based on the northern Shanghai community chronic disease management system on the follow-up compliance and satisfaction of patients with atrial fibrillation after cryoablation.

DETAILED DESCRIPTION:
Influence of patient-reported outcome follow-up based on the northern Shanghai community chronic disease management system on the follow-up compliance and satisfaction of patients with atrial fibrillation after cryoablation.Among patients with left atrial fibrillation after cryoablation at several sites, 240 consecutive eligible patients were randomly assigned to routine follow-up (control) and PRO (test) for 12 months. Follow-up, comparison of postoperative follow-up compliance, satisfaction, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old;Symptomatic, paroxysmal atrial fibrillation with cryoablation；Ability to understand and sign informed consent；

Exclusion Criteria:

* none

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Paroxysmal, symptomatic atrial fibrillation patients undergoing cryoablation；
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
follow-up rate | 1-year
  From the beginning of the study to the end of the study (a total of 12 months), the number of patients who completed each follow-up visit was standardized as a percentage of the total number of patients

SECONDARY OUTCOMES:
Anxiety Scale Score | 1 year
  Anxiety Scale Score
Depression Scale Score | 1 year
  Depression Scale Score
Quality of Life Scale Score | 1 year
  Quality of Life Scale Score

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, PhD, Study Chair — Tongji University
Locations (1):
- Jun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No